CLINICAL TRIAL: NCT01046110
Title: A Trial Comparing Efficacy and Safety of NN1250 With Sitagliptin in Insulin Naive Subjects With Type 2 Diabetes (BEGIN™ : EARLY)
Brief Title: Comparison of NN1250 With Sitagliptin in Subjects With Type 2 Diabetes Never Treated With Insulin
Acronym: BEGIN™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3580; U1111-1111-7126 (Other: WHO)
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Results first posted 2015-11-18 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg OD (Experimental)
  Interventions: Drug: insulin degludec
- DPP-IV inhibitor (Experimental)
  Interventions: Drug: sitagliptin

INTERVENTIONS:
Drug: insulin degludec — Injected under the skin once daily for 26 weeks. The doses will be individually adjusted.
  Arms: IDeg OD
Drug: sitagliptin — Sitagliptin tablets administered orally once a day at the same time every day for 26 weeks
  Arms: DPP-IV inhibitor

SUMMARY:
This trial will be conducted in Africa, Asia, North America and South America. The aim of this clinical trial is to compare NN1250 (insulin degludec) with sitagliptin, as add-on to subject's own current oral antidiabetic (OAD) treatment, in subjects with type 2 diabetes inadequately controlled with 1-2 OADs (metformin, sulphonylurea, glinides or pioglitazone).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (diagnosed clinically) for at least 6 months
* Ongoing treatment with 1 or 2 of the following OADs (metformin, insulin secretagogue (sulphonylurea or glinides) or pioglitazone) in any combination with unchanged dosing for at least 3 months prior to Visit 1 with the minimum doses stated: -Metformin: alone or in combination (including fixed combination)1500 mg or maximum tolerated dose (at least 1000 mg daily) -Insulin secretagogue (sulfonylurea or glinide): minimum half of the maximal daily dose according to local labelling -Pioglitazone: minimum half of the maximal daily dose according to local labelling or maximum tolerated dose
* Body Mass Index (BMI) below or equal to 40.0 kg/m^2
* HbA1c 7.5-11.0 % (both inclusive) by central laboratory analysis

Exclusion Criteria:

* Use within the last 3 months prior to Visit 1 of: exenatide, liraglutide, rosiglitazone or acarbose
* Cardiovascular disease, within the last 6 months prior to Visit 1, defined as: stroke; decompensated heart failure New York Heart Association (NYHA) class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty
* Uncontrolled treated/untreated severe hypertension (systolic blood pressure at least 180 millimetre (mm) mercury (Hg) and/or diastolic blood pressure at least 100 mmHg)
* Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemic event during the last 12 months) or hypoglycaemic unawareness as judged by the Investigator or hospitalisation for diabetic ketoacidosis during the previous 6 months
* Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate
* Cancer and medical history hereof (except basal cell skin cancer or squamous cell skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (83):
- United States (51):
  - Novo Nordisk Investigational Site, Huntsville, Alabama
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Greenbrae, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Mission Hills, California
  - Novo Nordisk Investigational Site, Palm Springs, California
  - Novo Nordisk Investigational Site, Torrance, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Inverness, Florida
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Ocala, Florida
  - Novo Nordisk Investigational Site, Ponte Vedra, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Columbus, Georgia
  - Novo Nordisk Investigational Site, Decatur, Georgia
  - Novo Nordisk Investigational Site, Dunwoody, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Huntington, Indiana
  - Novo Nordisk Investigational Site, Council Bluffs, Iowa
  - Novo Nordisk Investigational Site, Des Moines, Iowa
  - Novo Nordisk Investigational Site, Paducah, Kentucky
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Brockton, Massachusetts
  - Novo Nordisk Investigational Site, Livonia, Michigan
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Saint Paul, Minnesota
  - Novo Nordisk Investigational Site, Jackson, Mississippi
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, New Hyde Park, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Durham, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Murrells Inlet, South Carolina
  - Novo Nordisk Investigational Site, Corpus Christi, Texas
  - Novo Nordisk Investigational Site, El Paso, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Tomball, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Virginia Beach, Virginia
  - Novo Nordisk Investigational Site, Spokane, Washington
- Argentina (6):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, Caba
  - Novo Nordisk Investigational Site, Ciudad Autónoma de BsAs
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Mar del Plata
  - Novo Nordisk Investigational Site, Mendoza
- Canada (10):
  - Novo Nordisk Investigational Site, Surrey, British Columbia
  - Novo Nordisk Investigational Site, Cambridge, Ontario
  - Novo Nordisk Investigational Site, Chatham, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Smiths Falls, Ontario
  - Novo Nordisk Investigational Site, St. Catharines, Ontario
  - Novo Nordisk Investigational Site, Gatineau, Quebec
  - Novo Nordisk Investigational Site, Laval, Quebec
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, Saint-Marc-des-Carrieres, Quebec
- India (7):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Madurai, Tamil Nadu
  - Novo Nordisk Investigational Site, Nagpur
  - Novo Nordisk Investigational Site, Pune
- Mexico (2):
  - Novo Nordisk Investigational Site, Guadalajara
  - Novo Nordisk Investigational Site, Mexico City
- South Africa (3):
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
  - Novo Nordisk Investigational Site, Umhlanga
- Turkey (Türkiye) (4):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Denizli
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Izmir

REFERENCES:
- [Result] Philis-Tsimikas A, Del Prato S, Satman I, Bhargava A, Dharmalingam M, Skjoth TV, Rasmussen S, Garber AJ. Effect of insulin degludec versus sitagliptin in patients with type 2 diabetes uncontrolled on oral antidiabetic agents. Diabetes Obes Metab. 2013 Aug;15(8):760-6. doi: 10.1111/dom.12115. Epub 2013 May 6. PMID 23577643
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 78 sites in 7 countries: Argentina (2 sites), Canada (11 sites), India (8 sites), Mexico (2 sites), South Africa (3 sites), Turkey (5 sites) and the United States (47 sites).
Groups:
- IDeg OD: Insulin degludec (IDeg) was given once daily subcutaneously (s.c.) for 26 weeks with pre-trial treatment being 1 or 2 oral anti-diabetic drugs (metformin, sulfonylureas, glinides, pioglitazone) in any combination. Variation in injection time from day to day was allowed (minimum 8 hours and maximum 40 hours between injections).
- DPP-IV Inhibitor: Sitagliptin was given once daily dose of 100 mg for 26 weeks with pre-trial treatment being 1 or 2 oral anti-diabetic drugs (metformin, sulfonylureas, glinides, pioglitazone) in any combination.
Period: Overall Study
Arm/Group | IDeg OD | DPP-IV Inhibitor
Started | 229 | 229
Exposed | 226 (2 subjects were randomised in error and 1 subject did not want to take insulin) | 228 (1 subject was randomised in error)
Completed | 174 | 174
Not Completed | 55 | 55
Not completed — Adverse Event | 9 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 7 | 12
Not completed — Withdrawal Criteria | 3 | 5
Not completed — Unclassified | 36 | 35

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomised patients except for 11 subjects whose site was closed (4 subjects with IDeg; 7 subjects with DPP-IV group/arm). For 4 subjects each in IDeg OD and DPP-IV inhibitor arm, the fasting plasma glucose (FPG) values were missing at baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg OD | DPP-IV Inhibitor | Total
Number analyzed (Participants) | 225 | 222 | 447
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (10.2) | 54.9 (11.4) | 55.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 101 | 185
  Male | 141 | 121 | 262
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.8 (1.0) | 9.0 (1.0) | 8.9 (1.0)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 9.4 (2.6) | 9.9 (3.1) | 9.7 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline in HbA1c after 26 weeks of treatment
Time Frame: Week 0, Week 26
Population: The full analysis set (FAS) included all randomised subjects and missing data was imputed using last observation carried forward (LOCF). A site was closed, hence 11 randomised subjects (4 subjects with IDeg; 7 subjects with DPP-IV group/arm) were excluded from the FAS.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg OD | DPP-IV Inhibitor
Number analyzed (Participants) | 225 | 222
percentage of glycosylated haemoglobin | -1.56 (1.09) | -1.22 (1.16)

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change from baseline in FPG after 26 weeks of treatment
Time Frame: Week 0, Week 26
Population: The FAS included all randomised subjects and missing data was imputed using LOCF. One site was closed, hence 11 randomised subjects (4 in IDeg and 7 in DPP-IV group/arm) were excluded from the FAS. Fasting plasma glucose values were missing for another 8 subjects, hence did not contribute to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg OD | DPP-IV Inhibitor
Number analyzed (Participants) | 221 | 218
mmol/L | -3.22 (3.17) | -1.39 (3.11)

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 26 weeks + 7 days follow-up
Description: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDeg OD | DPP-IV Inhibitor
Serious Adverse Events (participants affected / at risk) | 14/226 | 10/228
Other Adverse Events (participants affected / at risk) | 44/226 | 53/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD (N=226) | DPP-IV Inhibitor (N=228)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Fallopian tube cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD (N=226) | DPP-IV Inhibitor (N=228)
Diarrhoea (Gastrointestinal disorders) | 13 (29) | 19 (27)
Nausea (Gastrointestinal disorders) | 8 (8) | 14 (14)
Nasopharyngitis (Infections and infestations) | 13 (14) | 18 (22)
Headache (Nervous system disorders) | 24 (38) | 15 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.